CLINICAL TRIAL: NCT03706638
Title: Daily vs. Intermittent Iron Therapy in Iron Deficient Pregnant Patients: A Randomized Noninferiority Trial
Brief Title: Daily vs Intermittent Iron Therapy in Pregnancy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: UConn Health (Other)
Responsible Party: Principal Investigator, Winston Campbell, Professor, Obstetrics and Gynecology; Maternal Fetal Medicine Fellowship Program Director, UConn Health
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 18-181-1
Record Dates: First submitted 2018-10-11; First posted 2018-10-16 (Actual); Last update posted 2020-04-21 (Actual); Status verified 2020-04

CONDITIONS: Iron Deficiency Anemia of Pregnancy
Keywords: Iron Deficiency Anemia; Pregnancy; Side Effects
MeSH Terms: conditions — Anemia, Iron-Deficiency | interventions — ferrous sulfate

STUDY DESIGN:
Intervention Model Description: Randomized Noninferiority Trial
Masking Description: Treatment groups are blinded and becomes unmasked when assigning the patient to a treatment group. At this time, the patient and the investigator becomes aware of the treatment assigned.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Daily (Other): Patients randomized to this arm will take ferrous sulfate 325 mg every day.
  Interventions: Dietary Supplement: Ferrous Sulfate
- Intermittent (Every other day) (Other): Patient's randomized to this arm will take ferrous sulfate 325 mg every other day.
  Interventions: Dietary Supplement: Ferrous Sulfate

INTERVENTIONS:
Dietary Supplement: Ferrous Sulfate — Patients would be randomized to either taking ferrous sulfate daily or every other day (on non consecutive days).

SUMMARY:
This is a randomized non inferiority trial to evaluate the response to iron therapy in the standard daily vs. intermittent (three-four times a week on nonconsecutive days) groups by using hematological markers (hemoglobin, hematocrit, transferrin, hepcidin, ferritin, human soluble transferrin receptor). The secondary outcome is to evaluate gastrointestinal discomfort and adherence to therapy between two treatment groups.

DETAILED DESCRIPTION:
The Centers for Disease Control and Prevention estimates that as many as 8 million American women of childbearing age are iron deficient. In a typical singleton gestation, the maternal need for iron averages close to 1000 mg. Of this 300 mg is for the fetus and placenta; 500 mg for maternal hemoglobin mass expansion; and 200 mg that is normally shed through the gut, urine, and skin. The total amount of 1000 mg considerably exceeds the iron stores of most women and results in iron-deficiency anemia unless iron supplementation is given.

Correction of anemia and restitution of iron stores can be accomplished with simple iron compounds-ferrous sulfate, fumarate or gluconate. Oral iron is an effective treatment for iron deficiency anemia and is inexpensive, safe and widely available.

In the past, a standard approach to the treatment of iron deficiency anemia was oral ferrous sulfate 325 mg (65 mg elemental iron) spaced in 3 doses each day for a total daily dose of 195 mg elemental iron. However, recent absorption studies concluded that maximal absorption of iron occurs with a dose in the range of 40 to 80 mg of elemental iron daily. This study was done in non pregnant iron-deficient women. Greater doses do not result in more iron absorption and are associated with more side effects. The findings of this study have been implemented by many into various areas of medicine.

Daily oral supplementation in pregnant women has been a long-standing, cost-effective recommended intervention both in the public health and clinical fields. However, adherence to daily iron and folic acid supplementation still faces challenges. Data from national surveys from 46 countries (2003 to 2009) indicate that about 52% to 75% of mothers receive any iron tablets during pregnancy, and the duration of supplementation is usually short.

According to a study by Khalafallah, the side effects or oral iron therapy including gastrointestinal disturbances characterized by colicky pain, nausea, vomiting, diarrhea, and constipation occur in about 50% of a patient taking iron preparations, and the investigators estimate that their patients have similar complaints and intolerances.

Many pregnant women taking oral iron, especially at doses greater than 30 mg daily of elemental iron daily, have gastrointestinal side effects, which cause them to discontinue the iron therapy. Taking iron supplementation on an intermittent basis may help to reduce gastrointestinal side effects and improve iron stores.

In the United States, the oral iron preparation of ferrous sulfate is often used to replete iron-deficient women. To the investigators' knowledge, studies have not been performed to evaluate daily vs. oral intermittent oral iron therapy in the United States, which has a different nutritional status and access to health care than other countries.

This study will randomize patients to the standard therapy: taking iron ferrous sulfate 325 mg (daily) by mouth once a day by mouth or intermittent therapy of taking ferrous sulfate 325 mg three- four times a week on alternating days. Hematological markers (hemoglobin, hematocrit, transferrin, hepcidin, ferritin, human soluble transferrin receptor), will be assessed prior to treatment and after treatment is completed.

ELIGIBILITY:
Inclusion Criteria:

1. Pregnant women who are not underweight (BMI < 18.5 kg/m2)
2. Reproductive-aged women 18-50
3. Singleton Pregnancy.
4. Patients undergoing third trimester blood work from 26-28 weeks.
5. Women who have had previously normal first-trimester blood work (hemoglobin, hematocrit, MCV) without any evidence of existing anemia.
6. Pregnant women with anemia designated with hemoglobin concentration less than 11 g/dL or hematocrit less than 33%
7. No pre-existing iron deficiency anemia or not already on iron supplementation.

Exclusion Criteria:

1. Women with medical problems known to affect iron metabolism or homeostasis
2. Women with existing thalassemias or anemias.
3. Women with abnormal bloodwork indicating anemia earlier in the pregnancy.
4. Women are already taking iron supplementation during the pregnancy for treatment of iron deficiency anemia.
5. Chronic illness is influencing iron absorption.
6. Underlying malabsorption disease.
7. History of bariatric surgery.
8. Severe anemia with maternal hemoglobin levels less than 6 g/dL
9. Preterm Labor, PPROM, signs of infection.

Ages: 18 Years to 50 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 46 (Actual)
Dates: Start 2018-10-25 (Actual); Primary Completion 2020-03-23 (Actual); Study Completion 2020-03-23 (Actual)

PRIMARY OUTCOMES:
Hematologic values assessed for anemia | This will be measured 4-6 weeks after starting treatment.
  Hematologic values of hemoglobin, hematocrit, transferrin, hepcidin, human soluble transferrin receptor and ferritin.

SECONDARY OUTCOMES:
Scores on self report survey of gastrointestinal adverse side effects after oral iron supplementation | Side effects will be reviewed every 2 weeks for a period of 4-6 weeks.
  The study adapts a previously validated questionnaire to capture side effects normally associated with oral iron supplementation. A likert scale is used with intermediate anchors to quantify side effects as absent, mild, moderate or severe. Absent was 0 symptoms experienced. Mild was less than 3 times a week, moderate was 3-5 times a week and severe was every single day. The possible total score is 60 with higher numbers representing more severe symptoms. These numbers will be compared between the two treatment groups.

CONTACTS AND LOCATIONS:
Locations (1):
- UConn Health, Farmington, Connecticut, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Looker AC, Dallman PR, Carroll MD, Gunter EW, Johnson CL. Prevalence of iron deficiency in the United States. JAMA. 1997 Mar 26;277(12):973-6. doi: 10.1001/jama.1997.03540360041028. PMID 9091669
- [Background] American College of Obstetricians and Gynecologists. ACOG Practice Bulletin No. 95: anemia in pregnancy. Obstet Gynecol. 2008 Jul;112(1):201-7. doi: 10.1097/AOG.0b013e3181809c0d. Erratum In: Obstet Gynecol. 2020 Jan;135(1):222. doi: 10.1097/AOG.0000000000003624. PMID 18591330
- [Background] Khalafallah AA, Dennis AE. Iron deficiency anaemia in pregnancy and postpartum: pathophysiology and effect of oral versus intravenous iron therapy. J Pregnancy. 2012;2012:630519. doi: 10.1155/2012/630519. Epub 2012 Jun 26. PMID 22792466
- [Background] Daru J, Allotey J, Pena-Rosas JP, Khan KS. Serum ferritin thresholds for the diagnosis of iron deficiency in pregnancy: a systematic review. Transfus Med. 2017 Jun;27(3):167-174. doi: 10.1111/tme.12408. Epub 2017 Apr 20. PMID 28425182
- [Background] van den Broek NR, Letsky EA, White SA, Shenkin A. Iron status in pregnant women: which measurements are valid? Br J Haematol. 1998 Dec;103(3):817-24. doi: 10.1046/j.1365-2141.1998.01035.x. PMID 9858238
- [Background] Koenig MD, Tussing-Humphreys L, Day J, Cadwell B, Nemeth E. Hepcidin and iron homeostasis during pregnancy. Nutrients. 2014 Aug 4;6(8):3062-83. doi: 10.3390/nu6083062. PMID 25093277
- [Background] Cook JD, Flowers CH, Skikne BS. The quantitative assessment of body iron. Blood. 2003 May 1;101(9):3359-64. doi: 10.1182/blood-2002-10-3071. Epub 2003 Jan 9. PMID 12521995
- [Background] Stoffel NU, Cercamondi CI, Brittenham G, Zeder C, Geurts-Moespot AJ, Swinkels DW, Moretti D, Zimmermann MB. Iron absorption from oral iron supplements given on consecutive versus alternate days and as single morning doses versus twice-daily split dosing in iron-depleted women: two open-label, randomised controlled trials. Lancet Haematol. 2017 Nov;4(11):e524-e533. doi: 10.1016/S2352-3026(17)30182-5. Epub 2017 Oct 9. PMID 29032957
- [Result] F. Gary Cunningham, John C. Hauth, Kenneth J. Leveno, Larry Gilstrap Iii, Steven L. Bloom, & Katharine D. Wenstrom. (2010). Williams obstetrics. Williams Obstetrics (pp. 1081).
- [Result] Pena-Rosas JP, De-Regil LM, Dowswell T, Viteri FE. Intermittent oral iron supplementation during pregnancy. Cochrane Database Syst Rev. 2012 Jul 11;7(7):CD009997. doi: 10.1002/14651858.CD009997. PMID 22786531
- [Result] Tolkien Z, Stecher L, Mander AP, Pereira DI, Powell JJ. Ferrous sulfate supplementation causes significant gastrointestinal side-effects in adults: a systematic review and meta-analysis. PLoS One. 2015 Feb 20;10(2):e0117383. doi: 10.1371/journal.pone.0117383. eCollection 2015. PMID 25700159